CLINICAL TRIAL: NCT05907707
Title: Effects of Transcranial Alternating Current Stimulation (tACS) at Gamma Band Frequencies on Memory Recall and Sleep in Healthy Elderly Participants
Brief Title: Effects of Gamma-tACS on Memory and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 23-0597
Record Dates: First submitted 2023-05-18; First posted 2023-06-18 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-11

CONDITIONS: Transcranial Alternating Current Stimulation; Aging; Cognitive Decline; Memory; Sleep
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- First gamma (40Hz) stimulation, then active control (21Hz) stimulation (Experimental): After collecting sleep EEG at home for one night to acclimate to the data collection during sleep, participants first receive gamma (40Hz) tACS on Day 1 followed by a 5-9 day washout. Participants then receive active control (21Hz) stimulation.
  Interventions: Device: Gamma transcranial alternating current stimulation; Device: Control transcranial alternating current stimulation; Device: EEG headband; Device: Actigraphy wristband
- First active control (21 Hz) stimulation, then gamma (40 Hz) stimulation (Experimental): After collecting sleep EEG at home for one night to acclimate to the data collection during sleep, participants first receive active control (21Hz) tACS on Day 1 followed by a 5-9 day washout. Participants then receive gamma (40Hz) stimulation.
  Interventions: Device: Gamma transcranial alternating current stimulation; Device: Control transcranial alternating current stimulation; Device: EEG headband; Device: Actigraphy wristband

INTERVENTIONS:
Device: Gamma transcranial alternating current stimulation — tACS (gamma frequency, 40Hz) during cognitive testing (about 40 minutes duration).
  Other Names: DC-STIMULATOR MC Stimulator Plus
Device: Control transcranial alternating current stimulation — tACS (control frequency, 21Hz) during cognitive testing (about 40 minutes duration).
  Other Names: DC-STIMULATOR MC Stimulator Plus
Device: EEG headband — At-home, ambulatory, single-channel EEG headband which records brain activity during sleep
  Other Names: ULTEEMNite
Device: Actigraphy wristband — At-home, ambulatory, wrist-worn accelerometer which records levels of motor activity during the whole day

SUMMARY:
The purpose of this clinical trial is to investigate the feasibility and efficacy of non-invasive transcranial alternating current stimulation (tACS) at gamma frequency in enhancing memory recall and modulating sleep network dynamics measured by at-home electroencephalography (EEG) in healthy elderly people. Eligible participants will first collect sleep EEG at home for one night to acclimate to the data collection during sleep. Participants are then randomized into first undergoing either tACS at gamma band frequencies (i.e. 40Hz) or tACS at a control frequency (i.e. 21Hz). Stimulation is administered in the lab during a cognitive testing battery that includes memorizing items. After a night of sleep with EEG at home, participants return to the lab the following day to measure memory recall. Recall is performed again after five days. This sequence of encoding during stimulation in the lab, sleep EEG at home for one night, and recall is then repeated for the other stimulation condition about a week later. Participants are wearing an actigraphy wristband throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* >50 years old

Exclusion Criteria:

* Implanted device or metal in head (including cochlear implant or other hearing aid), cardiac pacemaker or any other powered medical device
* Known neurological disease from history (epilepsy, sleep disorder (insomnia, sleep apnea, restless legs syndrome, parasomnia), stroke or transitory ischemic attack, cognitive impairment, neurodegenerative disease (for example Alzheimer's disease, Parkinson's disease or amyotrophic lateral sclerosis), immune-mediated disease of the central nervous system, chronic infectious brain disease, brain tumor, traumatic brain injury with loss of consciousness and/or intracranial bleeding, chronic pain with the need for daily analgesic use)
* Positive screening for epilepsy (questionnaire)
* Pathological Montreal Cognitive Assessment (MoCA <26/30 points)
* Brain surgery in the past (lifetime)
* Known psychiatric disorder from history (schizophrenia (lifetime), obsessive compulsive disorder (OCD; lifetime), borderline personality disorder (lifetime), anxiety disorder (lifetime), bipolar disorder (lifetime), psychosis (lifetime), eating disorder (lifetime), depression (within the last three months)
* Positive screening for anxiety disorder (GAD-7 ≥10/21 points) or positive screening for depression (PHQ-9 ≥5/27 points)
* Known other relevant medical condition from history (moderate to severe chronic obstructive pulmonary disease (COPD), abnormal kidney function (defined as estimated Glomerular Filtration Rate <60ml/min), current liver disease (defined as hepatitis and/or liver cirrhosis), cancer, diabetes mellitus, cardiac disease (heart failure, myocardial infarct, atrial fibrillation and revascularization - all within the last three months)
* Working in night shifts or going to bed after midnight on 3 or more nights per week
* Positive screening for sleep disorder (PSQI >5/21 points)
* Psychotropic treatment or illegal drugs (including cannabis) within the last three months
* Indication for alcohol use disorder: AUDIT score (Alcohol Use Disorders Identification Test; screening for unhealthy alcohol use) ≥7 for females and for males ≥ 65 years or ≥8 for males <65 years
* Not willing to abstain alcohol at least 24 hours before each study visit
* Pregnancy, planned pregnancy, fertility treatment planned or ongoing
* Having experienced an adverse event in the past after receiving Transcranial Magnetic Stimulation (TMS)
* If, after filling out a questionnaire on the participant's medical history that informs researchers of relevant events that marginally increase the risk of an adverse event occurring during TMS, researchers will exercise their expert judgement to determine whether that participant should be excluded

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Center for Neurostimulation, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | First Gamma (40Hz) Stimulation, Then Active Control (21Hz) Stimulation | First Active Control (21 Hz) Stimulation, Then Gamma (40 Hz) Stimulation
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Washout (9 Days)
Arm/Group | First Gamma (40Hz) Stimulation, Then Active Control (21Hz) Stimulation | First Active Control (21 Hz) Stimulation, Then Gamma (40 Hz) Stimulation
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | First Gamma (40Hz) Stimulation, Then Active Control (21Hz) Stimulation | First Active Control (21 Hz) Stimulation, Then Gamma (40 Hz) Stimulation
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants who received transcranial alternating current stimulation: tACS.
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Customized [Count of Participants; unit: Participants]
  >50 Years of Age | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Tolerating Cognitive Testing During tACS
Description: To establish acceptability of tACS combined with cognitive testing in healthy elderly participants and will be considered acceptable if at least >/= 80% of participants tolerate the procedure.
Time Frame: Baseline (Day 1)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Number; unit: percentage of participants
Groups:
- Gamma (40Hz) Stimulation: Participants who received gamma (40Hz) tACS
  Gamma transcranial alternating current stimulation: tACS (gamma frequency, 40Hz) during cognitive testing (about 40 minutes duration).
- Active Control (21 Hz) Stimulation: Participants who received (21Hz) tACS
  Control transcranial alternating current stimulation: tACS (control frequency, 21Hz) during cognitive testing (about 40 minutes duration).
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
percentage of participants | 100 | 100

2. Primary Outcome: Verbal Memory at Day 1
Description: Participants will memorize 15 words ("Rey Auditory Verbal Learning Test") during gamma-tACS or control-tACS. They will be required to recall the words on the same day. The number of correctly remembered words will be recorded.
Time Frame: Baseline (Day 1)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Mean (Standard Deviation); unit: Number of words recalled
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
Number of words recalled | 7.7 (1.7) | 6.9 (2.4)

3. Primary Outcome: Verbal Memory at Day 2
Description: Participants will memorize 15 words ("Rey Auditory Verbal Learning Test") during gamma-tACS or control-tACS. They will be required to recall the words on the day after. The number of correctly remembered words will be recorded.
Time Frame: Follow-Up (Day 2)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Mean (Standard Deviation); unit: Number of words recalled
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
Number of words recalled | 5.7 (1.9) | 5.5 (2.5)

4. Primary Outcome: Verbal Memory at Day 5
Description: Participants will memorize 15 words ("Rey Auditory Verbal Learning Test") during gamma-tACS or control-tACS. They will be required to recall the words after 5 days. The number of correctly remembered words will be recorded.
Time Frame: Follow-Up (Day 5)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Mean (Standard Deviation); unit: Number of words recalled
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
Number of words recalled | 4.1 (2.2) | 3.9 (2.3)

5. Primary Outcome: Associative Verbal Memory at Day 1
Description: Participants will memorize 8 word-pairs during gamma-tACS or control-tACS. They will be required to recall the pairs on the same day. The number of correctly remembered word pairs will be recorded.
Time Frame: Baseline (Day 1)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Mean (Standard Deviation); unit: Number of word pairs recalled
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
Number of word pairs recalled | 6.1 (0.6) | 5.7 (1.6)

6. Primary Outcome: Associative Verbal Memory at Day 2
Description: Participants will memorize 8 word-pairs during gamma-tACS or control-tACS. They will be required to recall the pairs on the day after. The number of correctly remembered word pairs will be recorded.
Time Frame: Follow-Up (Day 2)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Mean (Standard Deviation); unit: Number of word pairs recalled
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
Number of word pairs recalled | 5.9 (0.9) | 4.7 (1.9)

7. Primary Outcome: Associative Verbal Memory at Day 5
Description: Participants will memorize 8 word-pairs during gamma-tACS or control-tACS. They will be required to recall the pairs after 5 days. The number of correctly remembered word pairs will be recorded.
Time Frame: Follow-Up (Day 5)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Mean (Standard Deviation); unit: Number of word pairs recalled
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
Number of word pairs recalled | 5.9 (1.2) | 5.0 (1.7)

8. Primary Outcome: Percentage of Participants in Which it is Possible to Obtain at Least 4 Hours EEG Recording
Description: To establish feasibility of at-home use of a single-channel EEG device during sleep. This will be considered feasible if the device has been worn for at least 4 hours during the first night for >/= 80% of participants.
Time Frame: Baseline (Day 1)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Number; unit: percentage of participants
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
percentage of participants | 60 | 60

9. Primary Outcome: Percentage of Participants Who Wear the EEG Device During All Three Nights for at Least 4 Hours
Description: To establish acceptability of at-home use of the single-channel EEG device during multiple nights. Acceptability will be considered as given if the device has been worn for at least 4 hours during each of the three nights in >/=80% of participants.
Time Frame: Baseline (Day 1)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Number; unit: percentage of participants
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
percentage of participants | 10 | 10

10. Primary Outcome: Amount of Sleep Spindles in Sleep-EEG
Description: To investigate the effect of a single session of gamma-tACS (compared to control-tACS) on the number of sleep spindles occuring during the night after the intervention. Sleep spindles during the first two hours of sleep-EEG will be counted. A sleep spindle is defined as a train of sinusoidal waves with frequency 11-16 Hz and a duration of at least 0.5 seconds.
Time Frame: Baseline (Day 1)
Population: Data were not properly collected for some participants due to technical difficulties.
Measure: Mean (Standard Deviation); unit: Number of sleep spindles
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 5 | 5
Number of sleep spindles | 57.6 (116) | 35.8 (64.0)

11. Primary Outcome: Amount of Slow Wave Sleep in Sleep-EEG
Description: To investigate the effect of a single session of gamma-tACS (compared to control-tACS) on the amount of slow wave sleep (deep/delta sleep) occuring during the night after the intervention. The amount of slow wave sleep during the first two hours of sleep-EEG will be counted.
Time Frame: Baseline (Day 1)
Population: Data were not properly collected for some participants due to technical difficulties.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 5 | 5
minutes | 25.2 (31.2) | 23.2 (23.3)

12. Secondary Outcome: Performance in Phonematic Fluency-Correct Words
Description: To investigate the effect of a single session of gamma-tACS (compared to control-tACS) on a phonematic fluency-task during 1 minute. The number of correct words will be calculated.
Time Frame: Baseline (Day 1), Follow-Up (Day 2)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Mean (Standard Deviation); unit: Number of correct words
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
Number of correct words
  Baseline | 46.0 (13.3) | 45.5 (8.1)
  Follow-Up (Day 2) | 46.9 (10.8) | 47.8 (9.7)

13. Secondary Outcome: Performance in Phonematic Fluency-Perseverations
Description: To investigate the effect of a single session of gamma-tACS (compared to control-tACS) on a phonematic fluency-task (i.e. production of words that start with a specific letter) during 1 minute. Number of correct words, number of perseverations and number of rule breaks will be calculated.
Time Frame: Baseline (Day 1), Follow-Up (Day 2)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Mean (Standard Deviation); unit: number of perseverations
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
number of perseverations
  Baseline | 1.5 (2.1) | 1.1 (1.1)
  Follow-Up (Day 2) | 1.3 (1.1) | 1.1 (1.9)

14. Secondary Outcome: Performance in Phonematic Fluency-Rule Breaks
Description: To investigate the effect of a single session of gamma-tACS (compared to control-tACS) on a phonematic fluency-task during 1 minute. Number of correct words, number of perseverations and number of rule breaks will be calculated.
Time Frame: Baseline (Day 1), Follow-Up (Day 2)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Mean (Standard Deviation); unit: number of rule breaks
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
number of rule breaks
  Baseline | 0.9 (1.1) | 0.7 (1.3)
  Follow-Up (Day 2) | 2.0 (2.0) | 1.0 (1.3)

15. Secondary Outcome: Executive Functioning (Time to Complete Stroop Test)
Description: To investigate the effect of a single session of gamma-tACS (compared to control-tACS) on the Stroop Color and Word Test during and on the day after the intervention. Time for test completion and errors will be calculated. Selective attention was evaluated with the Stroop Color Word Interference Test. In the interference portion of this test, the subject identifies the color of ink in which words ("red", "green", or "blue") are printed, requiring the subject to inhibit their natural tendency to read the word. A subject's score is the time taken to identify 50 stimulus items. The time taken to complete the maze is inversely proportional to the cognitive function.
Time Frame: Baseline (Day 1), Follow-Up (Day 2)
Population: One participant was not exposed to 40 Hz due to their time constraints.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
seconds
  Baseline | 54.5 (7.2) | 58.6 (11.5)
  Follow-Up (Day 2) | 48.5 (6.6) | 53.2 (10.1)

16. Secondary Outcome: Executive Functioning (Trail Making Test)
Description: To investigate the effect of a single session of gamma-tACS (compared to control-tACS) on the Trail Making Test (TMT; connecting a set of numbers and numbers and letters as quickly as possible while maintaining accuracy) during and on the day after the intervention. The TMT (Part A and Part B) is a measure of visuomotor processing/sequencing speed. Participants must draw a line connecting numbers in ascending order as quickly as possible. Completion time in seconds is recorded (0-120, where lower scores represent better performance). Completion time of Part B is divided by completion time of Part A (Ratio B/A).
Time Frame: Baseline (Day 1), Follow-Up (Day 2)
Population: One participant was not exposed to 40 Hz due to their time constraints. Data were missing for another participant.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 9 | 9
ratio
  Baseline (Day 1) | 1.7 (0.6) | 1.9 (0.8)
  Follow-Up (Day 2) | 2.3 (0.9) | 1.9 (0.3)

17. Secondary Outcome: Attentional Performance (TAP)
Description: To investigate the effect of a single session of gamma-tACS (compared to control-tACS) on subtests of the Test of Attentional Performance (TAP) during and on the day after the intervention. Percentile ranks for the following subtests will be calculated: Alertness (reaction time under two conditions), Go/NoGo (stimuli that require a selective reaction, that is, to react or not to react), Divided Attention (a visual and an auditory task must be processed in parallel), Visual Scanning (a matrix-like arrangement of 5 x 5 stimuli is used, the aim being to detect whether this arrangement includes a critical stimulus or not).
Time Frame: Baseline (Day 1), Follow-Up (Day 2)
Population: Data are missing for some participants due to technical reasons resulting in data not being saved.
Measure: Mean (Standard Deviation); unit: percentile rank
Arm/Group | Gamma (40Hz) Stimulation | Active Control (21 Hz) Stimulation
Number analyzed (Participants) | 10 | 10
percentile rank
  Baseline (Day 1) Alertness | 31.4 (26.6) | 32.3 (26.0)
  Baseline (Day 1) Go/NoGo: number analyzed (Participants) | 9 | 9
  Baseline (Day 1) Go/NoGo | 42.8 (37.2) | 56.1 (26.7)
  Baseline (Day 1) Divided Attention Acoustic: number analyzed (Participants) | 9 | 9
  Baseline (Day 1) Divided Attention Acoustic | 26.2 (31.9) | 13.8 (16.2)
  Baseline (Day 1) Divided Attention Visual: number analyzed (Participants) | 9 | 9
  Baseline (Day 1) Divided Attention Visual | 42.6 (28.2) | 38.4 (28.1)
  Baseline (Day 1) Visual Scanning Critical | 65.0 (27.4) | 67.0 (24.5)
  Baseline (Day 1) Visual Scanning Non-Critical | 42.8 (27.2) | 39.0 (29.3)
  Follow-Up (Day 2) Alertness | 39.2 (29.9) | 36.2 (31.3)
  Follow-Up (Day 2) Go/NoGo: number analyzed (Participants) | 9 | 9
  Follow-Up (Day 2) Go/NoGo | 44.0 (31.5) | 47.6 (35.6)
  Follow-Up (Day 2) Divided Attention Acoustic: number analyzed (Participants) | 9 | 9
  Follow-Up (Day 2) Divided Attention Acoustic | 24.1 (25.0) | 19.0 (20.1)
  Follow-Up (Day 2) Divided Attention Visual: number analyzed (Participants) | 9 | 9
  Follow-Up (Day 2) Divided Attention Visual | 48.4 (28.6) | 57.3 (23.4)
  Follow-Up (Day 2) Visual Scanning Critical | 72.4 (29.0) | 72.0 (28.5)
  Follow-Up (Day 2) Visual Scanning Non-Critical | 47.8 (28.8) | 50.5 (28.7)

18. Other Pre Specified Outcome: Exploration of a Relationship (Correlation) Between the Amount of Sleep Spindles and Slow Wave Sleep With Recall
Description: A relationship is defined as a correlation (Pearson's) between memory recall performance (amount of words recalled) and sleep EEG features (especially spindles, slow waves), i.e., whether better memory recall is associated with more sleep spindles and more slow wave sleep in the night after stimulation.
Time Frame: Baseline (Day 1), Follow-Up (Day 2)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Exploration of a Relationship (Correlation) of Sleep-Wake-Schedule Changes and Type of Stimulation
Description: To see whether there is a correlation (Pearson's) between type of stimulation/wearing EEG and the motor activity pattern (measured by actigraphy wristband).
Time Frame: Baseline (Day 1), Follow-Up (Day 2)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the first intervention administration through follow-up, up to 14 days later.
Groups:
- First Gamma (40Hz) Stimulation: Participants who received gamma (40Hz) tACS
  Gamma transcranial alternating current stimulation: tACS (gamma frequency, 40Hz) during cognitive testing (about 40 minutes duration).
- First Active Control (21 Hz) Stimulation: Participants who received (21Hz) tACS
  Control transcranial alternating current stimulation: tACS (control frequency, 21Hz) during cognitive testing (about 40 minutes duration).
Arm/Group | First Gamma (40Hz) Stimulation | First Active Control (21 Hz) Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT05907707/Prot_SAP_000.pdf